CLINICAL TRIAL: NCT04186182
Title: The Child-In-Context-Intervention (CICI): The Feasibility of a Study Protocol for Treatment of Chronic Symptoms of Pediatric Acquired Brain Injury
Brief Title: Treating Chronic Symptoms of Pediatric Acquired Brain Injury - a Feasibility Study
Acronym: CICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: The Research Council of Norway (Other); Oslo University Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Monash University (Other); The Hospital of Vestfold (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunnaasRH
Record Dates: First submitted 2019-11-08; First posted 2019-12-04 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-10

CONDITIONS: Brain Injuries; Brain Diseases; Family; Child
Keywords: Rehabilitation
MeSH Terms: conditions — Brain Injuries; Brain Diseases

STUDY DESIGN:
Intervention Model Description: This is a feasibility trial evaluating the feasibility and acceptability of a planned randomized controlled trial. Therefore, no control group will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CICI - Feasibility trial study group (Other): The feasibility of the entire CICI-protocol will be evaluated. See details above.
  Interventions: Behavioral: CICI - Feasibility trial study group

INTERVENTIONS:
Behavioral: CICI - Feasibility trial study group — The intervention will include 7 individualized meetings with the family (2 home visits + 5 videoconferences), 2 parent group sessions and 4 meetings with school and local care providers, delivered over a 4-5 month period.
  Other Names: The CICI protocol

SUMMARY:
Children with acquired brain injury (ABI) often struggle with complex impairments, including cognitive (such as memory and attention), social, emotional and behavioral challenges. There is broad agreement that there is a lack of evidence-based knowledge about rehabilitation for children with ABI in the chronic phase. The current study is a feasibility study of a planned randomized controlled trial (RCT), the CICI-intervention, directed towards children with ABI and their families in the chronic phase. The feasibility study aims to evaluate the study protocol, the assessment procedures and the technical solutions prior to performing the RCT.

A feasibility study with six participating children and families will be conducted in close collaboration with schools and local health care providers. The intervention to be tested (the CICI-intervention) focuses on the child's and family's individually identified target outcome areas to be addressed, with corresponding rehabilitation goals. The intervention aims to enhance everyday functioning in the home and school environment by reducing ABI-related symptoms, and by attaining rehabilitation goals in areas noted as challenging by the participants. In the future RCT-study the efficacy of the CICI-intervention will be measured in terms of goal attainment, community participation, cognitive, behavioral, social, and family functioning.

DETAILED DESCRIPTION:
There is considerable knowledge about how to help children with ABI during the first, acute and post-acute stages. Yet, impairments are often long lasting and, due to the vulnerability of children's developing brain, new problems may emerge or become increasingly problematic over time. Children with ABI may struggle at school and with peers, which can lead to or increase emotional difficulties, and reduce quality of life, affecting the children and their families. The local communities and the children's schools are, together with the families, often left responsible for dealing with the chronic challenges of pABI. Parents may experience considerable stress and develop emotional symptoms when a child suffers an ABI. As a result, the entire family may experience impaired function, which in turn may affect the long-term prognosis of the child with ABI.

In this feasibility study, six children between 6 and 15 years will be included. The children will have a clinical ABI diagnosis, verified injury related intracranial abnormalities, and be more than one year post injury at inclusion. The child and/or their family must report enduring cognitive, emotional, social or physical challenges related to the brain injury. The intervention will be conducted in collaboration with the children's families, schools and their local care providers. It consists of individualized goal-oriented strategies adapted to the home- and school-setting. Goal attainment scaling will be applied. In addition, psychoeducation will be provided to the family and school/local care providers on topics related to the child's injury. Parent group sessions will be held for discussions and knowledge transfer concerning family challenges after a pABI, such as communication skills and parenting. The intervention will include 7 individualized meetings with the family (2 home visits + 5 videoconferences), 2 parent group sessions and 4 meetings with school and local care providers during a period of 4-5 months.

This feasibility study primarily aims to evaluate adherence to the CICI study protocol, responsiveness of participants and therapists, and the usefulness of the intervention. Furthermore, recruitment procedures, assessment protocol, goal setting and the technical solutions will be evaluated. A questionnaire developed for this project will be used to assess the families' satisfaction with the intervention as well as the acceptability of the intervention to families and therapists, while checklists, logs and qualitative interviews will be used to assess the remaining outcomes. Assessments in the future RCT will be conducted at baseline (T1), at the end of the intervention (T2, 4-5 months after inclusion) and one year after inclusion (T3). In the feasibility study, T1 and T2 will be included, as this is considered sufficient to evaluate feasibility of the study protocol as such.

The primary outcomes of the CICI-intervention in the future RCT-study, will be:

* severity of brain injury symptoms (Health and Behavior Inventory - HBI),
* the child's quality of life (The Pediatric Quality of Life Inventory - Peds-QL), and
* parenting self-efficacy (Tool to Measure Parenting Self-Efficacy - TOPSE/Teens TOPSE).

Secondary outcome measures of the CICI-intervention in the future RCT-study, will be:

* changes in self- and parental perceived severity of the individually defined target outcome areas (measured on a 5-point Likert scale),
* goal attainment scaling in the CICI group (Goal Attainment Scaling - GAS),
* emotional symptoms of the children (Child Behavior Checklist (CBCL), Teacher Report Form (TRF) and Youth Self-report (YSR))
* emotional symptoms of the parents (Patient Health Questionnaire 9 - PHQ-9 and Generalized Anxiety Disorder 7 - GAD-7),
* children's executive functioning in the home and school environment (Behavior Rating Inventory of Executive Function 2 - BRIEF-2),
* participation (The Child and Adolescent Scale of Participation - CASP),
* global outcome after pABI (Glasgow Outcome Scale Extended Pediatric Version - GOS-E Peds),
* parental stress (Parental Stress Scale - PSS)
* family functioning (Family Assessment Device - FAD), and
* unmet healthcare needs of the family (The Family Needs Questionnaire - Pediatric version - FNQ-P).

In addition, the neuropsychological screening battery performed at baseline in the future RCT-study will consist of the following test measures: Similarities, Matrix Reasoning, Coding, Digit Span from the Wechsler Intelligence Scale for Children-V, Inhibition and Comprehension of Instructions from Nepsy-II, the Children's Communication Checklist-2 questionnaire and the Children's Auditory Verbal Learning Test-2.

October 27, 2020: This feasibility study was recruiting and in early stages when the Covid-19 pandemic forced a halt in the study in March 2020. The insecurity of the situation caused us not to register the study as suspended, as we hoped from week to week that we would be able to continue. However, the pandemic resulted in a total halt, and reopening of the entire study in august 2020. The new timeline has been adjusted accordingly in the clinical trials.gov records.

ELIGIBILITY:
Inclusion Criteria:

* School-aged (6-15 years) children with clinical ABI-diagnosis and CT/MRI verified injury-related intracranial abnormalities, 1 year or more after injury. We anticipate including patients with the following etiologies: TBI, cerebrovascular incidents, anoxia, encephalitis and non-progressive brain tumors.
* The above-mentioned children, and/or their parents, report ABI-related cognitive, emotional, or behavioral problems that affect participation in activities with family, friends, school and/or community.
* The children attend school regularly, with or without injury-related adaptations.
* The family is able and willing to actively participate in a goal-oriented approach

Exclusion Criteria:

* Patients with severe pre- or comorbid neurological or neuropsychiatric disorders that would confound assessment and/or treatment outcomes.
* Patients with brain tumors in active treatment or at great risk of relapse.
* Patients with severe psychiatric illness or children with injuries so severe that they are in institutionalized care.
* Children in custody of the child protection services.
* Parental severe psychiatric illness, drug abuse or indications of a history of or risk of domestic violence.
* The family is not fluent in Norwegian

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Protocol adherence assessed by study-specific checklists | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The therapists will monitor discrepancies between intervention delivery and the CICI-manual by using extensive checklists relating to each of the intervention sessions. The number of non-delivered treatment components will be counted, and the percentage of deviation will be calculated compared to the total number of treatment components.
  High feasibility: 15 % deviation or less, Moderate feasibility: 15-25 % deviation, Low feasibility: > 25 % deviation
Child Responsiveness to the intervention assessed by ratings on the study specific Acceptability Scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The total mean score on the Responsiveness subscale (6 items) on the Acceptability Scale, rated by the child, will determine child responsiveness. The responsiveness subscale consists of the following items (the wording adapted to the child's age): I would recommend participating in the study to others, the therapist was warm and understanding, I trusted the therapist, I had the opportunity to state my opinions about the therapist's suggestions, my opinions were taken seriously, I was given sufficient information during the study about the work we were doing.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
Caregiver Responsiveness to the intervention assessed by ratings on the study specific Acceptability Scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The total mean score on the Responsiveness subscale (6 items) on the Acceptability Scale, rated by the caregiver, will determine caregiver responsiveness. The responsiveness subscale consists if the following items: I would recommend participating in the study to others, the therapist was warm and understanding, I trusted the therapist, I had the opportunity to state my opinions about the therapist's suggestions, my opinions were taken seriously, I was given sufficient information during the study about the work we were doing.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
a. Usefulness of the intervention assessed by child ratings on the study-specific Acceptability Scale for this study | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The total mean score on the Usefulness subscale (6 items) in the Acceptability Scale will determine perceived usefulness of the intervention. The child version of the usefulness subscale consists of the following items: The program has helped me, the program has helped my family, I would recommend participating in the program to others, I have learned something new that helps me, I have learned more about what I struggle with after the injury, I have learned what I can say to others about what I struggle with due to the injury.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
b. Usefulness of the intervention assessed by caregiver ratings on the study-specific Acceptability Scale for this study. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The total mean score on the Usefulness subscale (9 items) in the Acceptability Scale will determine perceived usefulness of the intervention. The caregiver version of the usefulness subscale consists of the following items:
  The program has helped my child, the program has helped my family, the program has helped me, I would recommend participating in the program to others, I have gained more insight into my child´s challenges, I will use my new knowledge in the future, I have used my new knowledge in other settings, I found it useful to meet other families who are in a similar situation as we are, the school meetings were useful.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.

SECONDARY OUTCOMES:
Recruitment procedures assessed by a) consent rate | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The therapist will log consent rate of families and schools. High feasibility: ≥ 30%, Moderate feasibility: 15-29%, Low feasibility: <15%
Recruitment procedures assessed by b) duration of phone calls and screening interview per family | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  Therapist will record duration of recruitment procedures, hereunder the telephone screening interview and other telephone calls. High feasibility: 3 hours or less, Moderate feasibility: ˃3 and ≤5 hours, Low feasibility: >5 hours
Recruitment procedures assessed by c) the number of participants excluded at or after baseline | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  High feasibility: One family excluded at or after baseline, Moderate feasibility: Two families excluded at or after baseline, Low feasibility: More than two families excluded at or after baseline
Recruitment procedures assessed by d) the number of families that completed the whole intervention | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  Description: Number of families out of six that participate in the first intervention meeting (after baseline) and complete the entire intervention.
  High feasibility: Six families completed the intervention, Moderate feasibility: Five families completed the intervention, Low feasibility: Four or fewer families completed the intervention
The burden of the assessment protocol for the child, reported by the child on the study-specific Acceptability Scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The total mean score on the following four items in the Acceptability Scale will determine the child burden of the assessment protocol: If the child was comfortable being tested and if the child was comfortable expressing his/her symptoms and opinions through the questionnaires, if the child understood the questionnaires and if the assessment made the child tired.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
The burden of the assessment protocol for the child, reported by caregivers on the study-specific Acceptability Scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The total mean score on the following four items in the Acceptability Scale will determine the child burden of the assessment protocol perceived by the caregiver: If the child was comfortable being tested, if the child was comfortable expressing his/her symptoms and opinions through the questionnaires, if the child understood the questionnaires and if the assessment made the child tired.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
The burden of the assessment protocol for the caregivers, reported by caregivers on the study-specific Acceptability Scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  Description: The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The following item in the Acceptability Scale will determine the caregiver burden of the assessment protocol: There were too many questionnaires.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
Caregiver reported relevance of topics in questionnaires | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The caregivers' perceived relevance of the topics in caregiver-questionnaires will be measured with two items on the Acceptability Scale: I was able to give important information through the questionnaires, the questionnaires were not relevant for me. Mean score will be calculated.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
Therapist reported burden of the baseline assessment measured by the duration of the assessment. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The therapist will record the duration of the baseline assessment through logs. High feasibility: ≤ 3hours, Moderate feasibility: ˃3 hours and ˂4 hours, Low feasibility: ≥4 hours
The perceived relevance of working with SMART-goals as rated by caregivers on the study-specific Acceptability Scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The perceived relevance of working with SMART-goals for the caregivers will be measured with three items on the Acceptability Scale ("The goals we set were important", "The strategies we used for working towards the goals have helped my family", "The strategies we used for working towards the goals have helped my child"). Mean score will be calculated.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
The perceived relevance of working with SMART-goals rated by the child on the study-specific Acceptability Scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree"). The perceived relevance of working with SMART-goals for the child will be measured with one item on the Acceptability Scale ("The goals we set were important").
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2.
Therapist-recorded technical failures in using videoconference in treatment delivery assessed by a study-specific log. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The therapist records the number of sessions interrupted due to technical failure, per family.
  High feasibility: Restart of equipment in 0-1 sessions per family, Moderate feasibility: Restart of equipment in 2-3 sessions per family, Low feasibility: Restart of equipment in 4-5 sessions per family.
Therapist-recorded time spent on installment of the equipment for using videoconference in treatment delivery | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The therapist will record the time spent on installing the technical equipment for video conference use, including software, per family.
  High feasibility: Installment completed in ≤ 20 minutes in one go, Moderate feasibility: Installment completed in > 20 minutes in one go, Low feasibility: Additional visit required to complete installment.
Experienced quality of communication in using videoconference in treatment delivery, assessed by the Acceptability scale. | Will be evaluated after the intervention period, i.e. 4-5 months after inclusion.
  The study-specific acceptability Scale is rated on a scale from 0 ("Completely disagree") to 4 ("Completely agree") and includes one question concerning the quality of communication through videoconference. The wording is adapted to the children's age, and the children, their parents, and the therapists will rate the question. The mean score will be calculated.
  High feasibility: Mean score ≥ 3 ("Agree"), Moderate feasibility: Mean score ≥ 2 and < 3, Low feasibility: < 2 on the item assessing quality of communication through videoconference.
Semi-structured qualitative interviews with all participating children, caregivers and teachers will be conducted to elaborate aspects of feasibility as described above. | Will be performed after the intervention period, i.e. 4-5 months after inclusion.
  Explored topics: responsiveness to the intervention, usefulness of the intervention, the perceived relevance of working with SMART-goals, and experienced quality of communication in using videoconference in treatment delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Løvstad, PhD, Principal Investigator — Sunnaas Rehabilitation Hospital, University of Oslo
Locations (1):
- Sunnaas rehabilitation hospital, Nesoddtangen, Norway

IPD SHARING:
Plan to Share IPD: No
Data are person sensitive and will not be openly shared.

REFERENCES:
- [Derived] Svendsen EJ, Killi EM, Rohrer-Baumgartner N, Holthe IL, Sandhaug M, Borgen IMH, Wade SL, Hauger SL, Lovstad M, Bragstad LK. Children's, parents', and teachers' experiences of the feasibility of a telerehabilitation intervention for children with acquired brain injury in the chronic phase - a qualitative study of acceptability and participation in the Child In Context Intervention (CICI). BMC Health Serv Res. 2023 Jun 8;23(1):603. doi: 10.1186/s12913-023-09589-z. PMID 37291543